CLINICAL TRIAL: NCT05578833
Title: Algorithm for Cervix Carcinoma Screening in the Czech Republic Using the Detection of HPV DNA With Selective HPV 16/18 Genotype and Special CINtec Plus Cytological Colouring
Brief Title: Algorithm for Cervix Carcinoma Screening in CZ Using the Detection of HPV DNA and CINtec Plus
Acronym: LIBUSE
Status: Completed | Type: Observational
Sponsor: AeskuLab Pathology Prague (Other)
Collaborators: Institute of Biostatistics and analyses, Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: IBA1132
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Algorithm for Cervix Carcinoma Screening
Keywords: HPV DNA; LIBUSE; CINtec plus; cytology; cervix carcinoma; human papilomavirus
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Human Papillomavirus DNA Tests; Genes, p16

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Smear from cervix
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: HPV DNA test with selective HPV 16/18 genotyping (cobas® 4800 HPV Test, Roche) — The enrolled patients underwent standard conventional cytology plus a test for the detection of high-risk human papilomavirus (hrHPV) with selective genotype specification (HPV 16, 18 and other hrHPV) - combined screening. In defined cases of positive hrHPV, the patient underwent reflexive examination by CINtec plus technology.
  After the initial combined screening the patients continued in the standard Czech screening practice (annual conventional cytology) or be treated according to the particular finding of the initial episode. For three years, the incidence of pre-cancers and invasive cervix carcinomas were monitored and data were entered into an electronic register.
  The second combined screening episode followed in year 3. An evaluation of its results immediately followed.
Diagnostic Test: p16 and Ki-67 biomarker detection in the form of dual cytological staining (CINtec Plus, Roche) — The enrolled patients underwent standard conventional cytology plus a test for the detection of high-risk human papilomavirus (hrHPV) with selective genotype specification (HPV 16, 18 and other hrHPV) - combined screening. In defined cases of positive hrHPV, the patient underwent reflexive examination by CINtec plus technology.
  After the initial combined screening the patients continued in the standard Czech screening practice (annual conventional cytology) or be treated according to the particular finding of the initial episode. For three years, the incidence of pre-cancers and invasive cervix carcinomas were monitored and data were entered into an electronic register.
  The second combined screening episode followed in year 3. An evaluation of its results immediately followed.
Diagnostic Test: standard conventional cytology PAP test — The enrolled patients underwent standard conventional cytology plus a test for the detection of high-risk human papilomavirus (hrHPV) with selective genotype specification (HPV 16, 18 and other hrHPV) - combined screening. In defined cases of positive hrHPV, the patient underwent reflexive examination by CINtec plus technology.
  After the initial combined screening the patients continued in the standard Czech screening practice (annual conventional cytology) or be treated according to the particular finding of the initial episode. For three years, the incidence of pre-cancers and invasive cervix carcinomas were monitored and data were entered into an electronic register.
  The second combined screening episode followed in year 3. An evaluation of its results immediately followed.

SUMMARY:
Cervix carcinoma has been a serious, long-term issue in the Czech Republic. The cause of nearly all cervix carcinomas is human papilomavirus (HPV). Hence the detection of the HPV genome is a more prospective screening tool with higher sensitivity than a cytological swab. As shown by comparative studies, the sensitivity of the HPV DNA test in the detection of severe pre-cancer is 35% higher on average when compared to the cytological test.

The study repeatedly determined the presence of the HPV genome, including the prevalence of selected HPV genotypes (16, 18 and other hrHPV) and conventional cytology. The relative sensitivity of the two methods was specified. In the course of the prospective follow-up, the incidence of pre-cancers and invasive tumours in the study population were specified.

DETAILED DESCRIPTION:
Cervix carcinoma has been a serious, long-term issue in the Czech Republic. About 1,000 new cases are diagnosed every year and about 400 female patients die as a result of the disease. More than 20,000 women in the Czech Republic live with a history of cervix carcinoma therapy and the potential risk of its recurrence. Although the past years have been marked with effective organisational changes in cervix carcinoma screening thanks to which a decreasing trend of its incidence can be observed, there is a lack of substantial impact on the occurrence of advanced stages of the disease and mortality. Similar data have also been reported internationally: foreign authors analysed cases of patients with a malignant cervix tumour. They reported that 24 - 32% of females with a diagnosed malignant tumour had periodically undergone cytological screening. The reason is that the sensitivity of an individual cytological examination for detecting severe pre-cancer is limited, ranging between 40 - 75% and only increasing with repeated examinations. The negative predictive value of the cytological swab is additionally limited and reaches 0.78% in recent studies over a three-year screening interval.

The cause of nearly all cervix carcinomas is human papilomavirus (HPV). Hence the detection of the HPV genome is a more prospective screening tool with higher sensitivity than a cytological swab. The sensitivity of the validated HPV DNA test using PCR method reaches 94.5% for detecting severe pre-cancer (confidence interval 94.2 - 96.9%). As shown by comparative studies, the sensitivity of the HPV DNA test for the detection of severe pre-cancer is 35% higher on average when compared to the cytological test. The HPV DNA test in addition shows a significantly better negative three-year predictive value (0.34%) and the low value continues for at least another five years. The lower specificity of the HPV DNA test can be compensated by selective genotype specification with proof of the most frequent oncogenic genotypes HPV 16 and HPV 18. This promising procedure, validated by large multicentric randomised studies and introduced to clinical practice in several European countries, primarily uses the detection of HPV DNA.

The study repeatedly determined the presence of the HPV genome, including the prevalence of selected HPV genotypes (16, 18 and other hrHPV) and conventional cytology. The relative sensitivity of the two methods was specified. In the course of the prospective follow-up, the incidence of pre-cancers and invasive tumours in the study population were specified.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signature
* Age 30 - 60
* Screening (not reviewing after previous abnormal cytological finding)
* Sampling of gravid women possible

Exclusion Criteria:

* Refusal to take part

Ages: 30 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Females 30 - 60 years
Sampling Method: Non-Probability Sample
Enrollment: 2426 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of hrHPV positivity in the Czech population | 49 months
  The ratio of patients with a positive HPV test in the first combined screening episode and the number of examined women.

SECONDARY OUTCOMES:
Specification of prevalence of selected hrHPV genotypes | 49 months
  Representation of individual hrHPV genotypes in the first and the second screening episode in all examined women and in all HPV positive women.
Detection level of pre-cancers and invasive carcinomas in the first combined screening episode (indicator of relative sensitivity of the two methods) | 49 months
  The ratio of detected diseases and the number of examined women in the first screening episode, a secondary endpoint.
Incidence of pre-cancers and invasive carcinomas in the course of the follow-up | 49 months
  The cumulative incidence of diseases considering the censored patients, a secondary endpoint.
Incidence of pre-cancers and invasive carcinomas after the second screening episode | 49 months
  The cumulative incidence of the disease in patients based on the initial HPV test results and initial cytology results.

CONTACTS AND LOCATIONS:
Overall Officials: Markéta Trnková, MD, Principal Investigator — Aeskulab Patologie, ks
Locations (1):
- Aeskulab Patologie, ks, Prague, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MJ, Castle PE, Lorincz AT, Wacholder S, Sherman M, Scott DR, Rush BB, Glass AG, Schiffman M. The elevated 10-year risk of cervical precancer and cancer in women with human papillomavirus (HPV) type 16 or 18 and the possible utility of type-specific HPV testing in clinical practice. J Natl Cancer Inst. 2005 Jul 20;97(14):1072-9. doi: 10.1093/jnci/dji187. PMID 16030305
- [Background] Kjaer SK, Frederiksen K, Munk C, Iftner T. Long-term absolute risk of cervical intraepithelial neoplasia grade 3 or worse following human papillomavirus infection: role of persistence. J Natl Cancer Inst. 2010 Oct 6;102(19):1478-88. doi: 10.1093/jnci/djq356. Epub 2010 Sep 14. PMID 20841605
- [Background] McMenamin M, McKenna M, McDowell A. Clinical Utility of CINtec PLUS Triage in Equivocal Cervical Cytology and Human Papillomavirus Primary Screening. Am J Clin Pathol. 2018 Oct 24;150(6):512-521. doi: 10.1093/ajcp/aqy073. PMID 30169728
- [Background] Meijer CJ, Berkhof J, Castle PE, Hesselink AT, Franco EL, Ronco G, Arbyn M, Bosch FX, Cuzick J, Dillner J, Heideman DA, Snijders PJ. Guidelines for human papillomavirus DNA test requirements for primary cervical cancer screening in women 30 years and older. Int J Cancer. 2009 Feb 1;124(3):516-20. doi: 10.1002/ijc.24010. PMID 18973271
- [Background] Petry KU, Schmidt D, Scherbring S, Luyten A, Reinecke-Luthge A, Bergeron C, Kommoss F, Loning T, Ordi J, Regauer S, Ridder R. Triaging Pap cytology negative, HPV positive cervical cancer screening results with p16/Ki-67 Dual-stained cytology. Gynecol Oncol. 2011 Jun 1;121(3):505-9. doi: 10.1016/j.ygyno.2011.02.033. Epub 2011 Mar 21. PMID 21420158
- [Background] Rijkaart DC, Berkhof J, Rozendaal L, van Kemenade FJ, Bulkmans NW, Heideman DA, Kenter GG, Cuzick J, Snijders PJ, Meijer CJ. Human papillomavirus testing for the detection of high-grade cervical intraepithelial neoplasia and cancer: final results of the POBASCAM randomised controlled trial. Lancet Oncol. 2012 Jan;13(1):78-88. doi: 10.1016/S1470-2045(11)70296-0. Epub 2011 Dec 14. PMID 22177579
- [Background] Ronco G, Dillner J, Elfstrom KM, Tunesi S, Snijders PJ, Arbyn M, Kitchener H, Segnan N, Gilham C, Giorgi-Rossi P, Berkhof J, Peto J, Meijer CJ; International HPV screening working group. Efficacy of HPV-based screening for prevention of invasive cervical cancer: follow-up of four European randomised controlled trials. Lancet. 2014 Feb 8;383(9916):524-32. doi: 10.1016/S0140-6736(13)62218-7. Epub 2013 Nov 3. PMID 24192252
- [Background] Sehnal B, Slama J. What next in cervical cancer screening? Ceska Gynekol. 2020 Winter;85(4):236-243. PMID 33562978
- [Background] Sheikh S, Biundo E, Courcier S, Damm O, Launay O, Maes E, Marcos C, Matthews S, Meijer C, Poscia A, Postma M, Saka O, Szucs T, Begg N. A report on the status of vaccination in Europe. Vaccine. 2018 Aug 9;36(33):4979-4992. doi: 10.1016/j.vaccine.2018.06.044. Epub 2018 Jul 4. PMID 30037416
- [Background] Whitlock EP, Vesco KK, Eder M, Lin JS, Senger CA, Burda BU. Liquid-based cytology and human papillomavirus testing to screen for cervical cancer: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2011 Nov 15;155(10):687-97, W214-5. doi: 10.7326/0003-4819-155-10-201111150-00376. Epub 2011 Oct 17. PMID 22006930
- [Background] Wright TC Jr, Behrens CM, Ranger-Moore J, Rehm S, Sharma A, Stoler MH, Ridder R. Triaging HPV-positive women with p16/Ki-67 dual-stained cytology: Results from a sub-study nested into the ATHENA trial. Gynecol Oncol. 2017 Jan;144(1):51-56. doi: 10.1016/j.ygyno.2016.10.031. Epub 2016 Oct 27. PMID 28094038
- [Background] Hajjar DP, Marcus AJ, Etingin OR. Platelet-neutrophil-smooth muscle cell interactions: lipoxygenase-derived mono- and dihydroxy acids activate cholesteryl ester hydrolysis by the cyclic AMP dependent protein kinase cascade. Biochemistry. 1989 Oct 31;28(22):8885-91. doi: 10.1021/bi00448a030. PMID 2557910
- [Result] Slama J, Dvorak V, Trnkova M, Skrivanek A, Hurdalkova K, Ovesna P, Novackova M. Importance of addition of HPV DNA testing to the cytology based cervical cancer screening and triage of findings with p16/Ki67 immunocytochemistry staining in 35 and 45 years old women LIBUSE trial data analysis. Ceska Gynekol. 2020 Winter;85(6):368-374. PMID 33711896
- [Derived] Slama J, Dvorak V, Trnkova M, Skrivanek A, Hrabcova K, Ovesna P, Novackova M. Is phased implementation of HPV testing and triage with dual staining the way to transform organized cytology screening? Eur J Cancer Prev. 2024 Mar 1;33(2):168-176. doi: 10.1097/CEJ.0000000000000844. Epub 2023 Sep 21. PMID 37751376